CLINICAL TRIAL: NCT06224972
Title: Usability and Performance Assessment of DormoTech VLAB
Brief Title: Evaluation of the Usability and Performance Assessment of the DormoTech VLAB Device as a Home Sleep Test
Status: Completed | Type: Observational
Sponsor: Dormotech Medical (Industry)
Collaborators: Assaf-Harofeh Medical Center (Other Government)
Responsible Party: Sponsor
Other Study IDs: VLAB_C_T_1
Record Dates: First submitted 2023-12-06; First posted 2024-01-25 (Actual); Last update posted 2024-01-25 (Actual); Status verified 2024-01

CONDITIONS: Sleep Disorder
Keywords: Sleep test; Sleep disorder; Home sleep tests; Physiological data recorder; Sleep diagnostics
MeSH Terms: conditions — Sleep Wake Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Observational group: The study is observational study - one group.
  Interventions: Device: Vlab

INTERVENTIONS:
Device: Vlab — The study is observational, there is no intervention.

SUMMARY:
The study is a comparative, self-controlled, randomized, prospective investigation designed to assess the usability and accuracy of the DormoTech Vlab and compare its performance with a full polysomnography (PSG) study conducted over one night in a sleep lab. For the purpose of this study, the selected PSG device used for comparison is the Nox A1 system (K192469). Participants were required to wear the DormoTech Vlab, answer questionnaires pre and post-study, and simultaneously undergo a full PSG test using the Nox system.

The statistical methodology for this study was designed to ensure a comprehensive analysis of the data, adhering to the standards set by the International Council for Harmonisation (ICH) E3 guideline

DETAILED DESCRIPTION:
The intended use of the V-Lab device is to serve as Type 2 Sleep test, an inexpensive, more comfortable device that can replace the full sleep study in a sleep lab and at-home environment.

The device is composed of three units, two of which are wearable and the third is a central unit responsible for communication; The head unit is worn on the face like a mask, and the body unit is a belt that is worn around the torso. After a few minutes of wearing the device, the patient will become ignorant of its presence. A small rechargeable 3V Li-ion battery operates both units.

The V-Lab system supports the connectivity of peripheral devices for capturing additional signals using Bluetooth technology, e.g. pulse oximeters. The V-Lab device collects and stores physiological signals such as EEG, EOG, EMG, Total Airflow, Snore, Respiratory Effort (Thoracic and Abdominal), Body and Head Position, and HR (derived from Plethysmography) Both the head and chest units communicate with the central units via Bluetooth, and the wearable units send the measured data to the central unit. The central unit receives the data, stores it within an internal flash drive, and transmits it via Wi-Fi to online servers for further diagnosis.

Using the recorded data, a physician can diagnose sleep disorders manually or use any sleep diagnostic system that supports EDF Formats.

The study Objectives are to assess the efficiency, usability, durability, safety, and patient satisfaction of the V-Lab device and to validate the level of agreement between the V-Lab device and a PSG.

The study's main outcome measures are patient feedback as determined by a satisfaction questionnaire, agreement and level of agreement between V-Lab and the referenced device (e.g. Bland-Altman plots of the mean versus the difference will be presented, and sensitivity and specificity analysis), and safety as defined by Adverse Events related to device use.

The study population will include patients seeking medical attention at a sleep clinic, age 22 years old and above and the subject is willing and able to comply with the requirements of the protocol, fully understands all elements of, and has signed and dated, the written informed consent form before initiation of protocol-specified procedures.

The exclusion criteria for the participants are subjects not willing to sign informed consent, subjects age is under 22 years old, subjects with implanted electronic devices of any kind, including cardiac pacemakers, or similar assistive devices, electronic infusion pumps, and implanted stimulators, subjects using exterior electronic devices of any kind during the procedure, such as TENS, or similar assistive devices, subjects with known allergies to device materials, subjects with irritated skin or open wound on the body at the site of device placement, and pregnant women.

Subjects will be recruited on two investigational sites: Shamir Medical Center- Be'er Ya'akov, Israel, and Millennium Sleep Clinic, Be'er Sheva, Israel, by the attending physician.

Subjects will go through a standard PSG monitoring which will be performed with a V-Lab device monitoring simultaneously in the sleep lab during one night.

The subject will be informed that participation in the study is voluntary, that he/she may withdraw from the study at any time and that withdrawal of consent will not affect his/her subsequent medical treatment (if any) or relationship with the treating physician. Subjects will be asked to fill out a satisfaction questionnaire and to report to the investigator Adverse Events.

Before studying active participation, the investigator will perform documentation of demography, relevant medical history, and medication consumption. The investigator will perform also a physical examination, including documentation of relevant medical and surgical history that may affect the experiment, based on the investigator's opinion (including precise diagnosis of disease) and Vital Signs (Pulse, Blood Pressure, Temperature). Steps will be taken to ensure the collected data are accurate, consistent, complete, and reliable.

ELIGIBILITY:
Inclusion criteria:

* Age of 22 years old and above.
* Willingness and ability to comply with the protocol requirements.
* Understanding and provision of signed and dated informed consent

Exclusion criteria:

* Unwillingness to sign informed consent.
* Age below 22 years.
* Presence of implanted electronic devices or use of exterior electronic devices during the procedure.
* Known allergies to device materials.
* Skin irritation or open wounds at the device placement site.
* Pregnancy.

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects were recruited in the sleep clinic by the attending physician, or sub-investigator.
  The participants were patients who were referred by physicians for a full sleep study at the sleep laboratory.
Sampling Method: Non-Probability Sample
Enrollment: 47 (Actual)
Dates: Start 2023-06-13 (Actual); Primary Completion 2023-08-12 (Actual); Study Completion 2023-08-12 (Actual)

PRIMARY OUTCOMES:
AHI Score and Classification | During night 1
  The AHI (apnea-hypopnea index) score was categorized and compared according to levels of severity:
  AHI = number of Apneas+Hypopneas/total sleep time
  Categorizing Normal <5, Mild: 5<AHI<15, Moderate: 15<AHI<30, Severe: 30<AHI

SECONDARY OUTCOMES:
Total Sleep Time (min) | During night 1
  Time from sleep onset to sleep offset (min)
Sleep Efficiency (%) | During night 1
  Total sleep time (min) / Total recorded time (min)
Sleep Stages (%) | During night 1
  Wake, N1, N2, N3, REM (% from total sleep time)
Sleep Latency (min) | During night 1
  Time to fall asleep from the record starting (min)
Wake After Sleep Onset (min) | During night 1
  The first wake after sleep onset (min)
REM Latency (min) | During night 1
  The amount of time elapsed between the onset of sleep to the first REM stage (min)
Total snore (%) | During night 1
  The number of snoring episodes divided by the hours of total sleep time
Body Position | During night 1
  Supine position, Left, Right, Up (% from Total Sleep Time)

OTHER OUTCOMES:
Usability Questionnaire | During night 1
  Usability was gauged using pre and post-study questionnaires, each utilizing a 5-point Likert scale. Descriptive statistics was employed to summarize the questionnaire results, with a focus on median scores and interquartile ranges. A score of 3 (Neutral) or higher should be achieved for at least 70% of the questions.
Safety Measures | During night 1
  The frequency and severity of adverse events (AEs).

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin D Fox, MD, Principal Investigator — Assaf-Harofeh Medical Center
Locations (1):
- Shamir Medical Center, Be’er Ya‘aqov, Israel

REFERENCES:
- [Derived] Fox BD, Shihab M, Nassir A, Kushinsky D, Barnea O, Tal A. Validation of a novel mask-based device for monitoring of comprehensive sleep parameters and sleep disordered breathing. Sleep Breath. 2025 Jan 20;29(1):83. doi: 10.1007/s11325-025-03250-1. PMID 39833613